CLINICAL TRIAL: NCT01257698
Title: A Prospective, Randomized Study Comparing the Effects of Topical Aqueous Suppressants on Intraocular Gas Duration Following Pars Plana Vitrectomy
Brief Title: Effect of Topical Aqueous Suppressants on Intraocular Gas Duration Following Pars Plana Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, Michele Formoso, Research Manager, Mid Atlantic Retina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-935
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Macular Hole; Retinal Detachment
Keywords: Vitrectomy; Gas bubble; Retinal detachment; Macular hole; Aqueous suppressant
MeSH Terms: conditions — Retinal Perforations; Retinal Detachment | interventions — dorzolamide; Timolol; Ophthalmic Solutions; dorzolamide-timolol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dorzolamide-timolol topical drops (Active Comparator)
  Interventions: Drug: Dorzolamide 2%-timolol 0.5% topical eyedrops
- Standard of care (No Intervention)

INTERVENTIONS:
Drug: Dorzolamide 2%-timolol 0.5% topical eyedrops — Dorzolamide 2%-timolol 0.5%, 1 drop in operated eye twice daily until gas bubble completely resorbed. Patients randomized to this arm are instructed to use this drop in addition to standard post-operative eye drops.
  Other Names: Cosopt
  Arms: Dorzolamide-timolol topical drops

SUMMARY:
The purpose of this study is to see if glaucoma eye drops (dorzolamide-timolol) have any effect on the duration of an intraocular gas bubble following pars plana vitrectomy.

DETAILED DESCRIPTION:
At the end of some retinal surgeries, a gas bubble is placed in the eye. In surgeries for retinal detachment, this gas bubble helps to keep the tear(s) in the retina sealed up while the eye is healing and prevent the retina from re-detaching. In macular hole surgeries (a defect in the center part of the retina), the gas bubble helps to seal up this hole in the center part of the retina. The gas bubble (sulfur hexafluoride) will slowly disappear from the eye over the course of approximately 2 weeks.

In some cases, the gas bubble disappears more quickly than the surgeon would wish. Several eye drops are currently available which help to lower the eye pressure in conditions such as glaucoma where the eye pressure is unacceptably elevated and is causing or may cause vision loss. These drops have been shown to keep the eye pressure controlled after surgery with injection of a gas bubble in the eye. However, little is known about the effect of these drops on the duration of the gas bubble. The goal of this study is to see if these glaucoma eye drops have any effect on the amount of time the gas bubble remains in the eye.

After surgery with a gas bubble (sulfur hexafluoride) is completed, patients will be randomly assigned (like a flip of a coin) to receive a glaucoma drop (dorzolamide-timolol) or no glaucoma drop. These drops are currently available from pharmacies with a prescription and are not "experimental." However, the use of these drops in this protocol is not to treat glaucoma but represents an "off-label" use. Patients assigned to receive a glaucoma drop will be provided with the medication. All patients will receive the standard post-operative drops regardless of which group they are assigned to. Patients will be taken care of before and after the surgery like any other patient undergoing this procedure. The investigators expect that you will be enrolled in this study for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for pars plana vitrectomy with intraocular gas tamponade with sulfur hexafluoride (e.g., retinal detachment, macular hole, other condition at the discretion of the investigator).
* Ability to provide written informed consent and comply with study assessments for the full duration of the study.

Exclusion Criteria:

* Prior trabeculectomy or tube shunt surgery.
* Current use of topical aqueous suppressants or other glaucoma medications.
* Aphakia or presence of anterior chamber intraocular lens implant.
* Known allergy or contraindication to sulfa or beta-blocker use (e.g., asthma, chronic obstructive pulmonary disease, bradycardia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Lee MS, Pasha M, Weitzman M. The effect of aqueous humor suppressants on intravitreal gas bubble duration in rabbits. Am J Ophthalmol. 1998 May;125(5):701-2. doi: 10.1016/s0002-9394(98)00006-3. PMID 9625556
- [Background] Mittra RA, Pollack JS, Dev S, Han DP, Mieler WF, Pulido JS, Connor TB. The use of topical aqueous suppressants in the prevention of postoperative intraocular pressure elevation after pars plana vitrectomy with long-acting gas tamponade. Ophthalmology. 2000 Mar;107(3):588-92. doi: 10.1016/s0161-6420(99)00083-4. PMID 10711900
- [Background] Benz MS, Escalona-Benz EM, Murray TG, Eifrig CW, Yoder DM, Moore JK, Schiffman JC. Immediate postoperative use of a topical agent to prevent intraocular pressure elevation after pars plana vitrectomy with gas tamponade. Arch Ophthalmol. 2004 May;122(5):705-9. doi: 10.1001/archopht.122.5.705. PMID 15136318
- [Result] Shah CP, Hsu J, Spirn MJ, Donoso L, Garg SJ. Topical aqueous suppression does not significantly affect duration of intraocular gas tamponade after vitrectomy. Retina. 2012 Jan;32(1):168-71. doi: 10.1097/IAE.0b013e31822092a4. PMID 21878847

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard post-operative drops
Period: Overall Study
Arm/Group | Dorzolamide-timolol Topical Drops | Standard of Care
Started | 12 | 9
Completed | 8 | 9
Not Completed | 4 | 0
Not completed — Protocol Violation | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorzolamide-timolol Topical Drops | Standard of Care | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 1 | 3 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Duration of Intraocular Gas
Description: Patients will self-monitor gas bubble duration and will receive weekly phone calls by the study coordinator until gas disappearance is confirmed.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dorzolamide-timolol Topical Drops | Standard of Care
Number analyzed (Participants) | 8 | 9
days | 17.1 (1.6) | 18.1 (2.4)

ADVERSE EVENTS:
Arm/Group | Dorzolamide-timolol Topical Drops | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes